CLINICAL TRIAL: NCT02309346
Title: A Randomized Clinical Trial Between Clindamycin Once and Thrice a Day in Septic Abortion.
Brief Title: Clindamycin Once a Day in Septic Abortion
Acronym: CLINDA-PRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0328
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Septic Abortion
Keywords: clindamycin; septic abortion
MeSH Terms: conditions — Abortion, Septic | interventions — Clindamycin

STUDY DESIGN:
Intervention Model Description: randomization in blocks of 4
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clindamycin once a day (Experimental): Clindamycin 2700mg+gentamycin 240mg+ 250ml sterile saline solution i.v. once a day until clinical improvement
  Interventions: Drug: Clindamycin
- clindamycin thrice a day (Active Comparator): Clindamycin 900mg i.v. 8/8 h diluted in 250ml of sterile saline solution. In one of the solutions, 240 mg of gentamicin was diluted once a day.
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Clindamycin — Use of Clindamycin 2700mg+gentamycin 240mg+ 250ml sterile saline solution i.v. once a day

SUMMARY:
Septic abortion is a serious condition. Women with septic abortion are treated with clindamycin plus gentamicin using divided doses, i.e., thrice a day.

The objective of this study is to compare the rates of cure between once or thrice a day use of clindamycin with gentamicin in cases of septic abortion.

DETAILED DESCRIPTION:
Obstetric infections are very common, especially in developing countries, as a consequence of the practice of unsafe abortion. In these countries, an estimated five million women each year are hospitalized due to complications from induced abortions, which equates to a rate of 5-7 per thousand women.

Abortion remains a leading cause of maternal death in developing countries. According to the World Health Organization, it is estimated that 1 in 8 maternal deaths occur from complications of illegal abortion. Septic abortions play an important role in the maternal morbidity and mortality. The diagnosis of septic abortion should be considered when a woman of reproductive age presents with menstrual delay, vaginal bleeding accompanied by abdominal pain and fever.

In 1989, Plaisance et al. demonstrated that Clindamycin, an antibiotic used for septic abortion, could be prescribed at a dose of 12/12 hours, and bacterial inhibitory serum levels were similar to those in divided doses 6/6 hours. In 2003, Livingston et al. published the results of gentamicin and clindamycin combined in a single daily dose for cases of post-cesarean endometritis. Administration of clindamycin differed by being in a dose of 2700mg daily dose of different fractional 6/6 hours, or 8/8 hours, and the cure rates were 82% (45 of 56 cases successes) in a single daily dose (13). The etiology of postpartum endometritis is similar to that in infected abortion (14, 15), but little information exists regarding the use of single daily dose in this disease.

A retrospective study recently conducted by our group showed that patients with infected abortion treated with Clindamycin single dose achieved cure rates of 98% (95% CI - 95 to 99%), suggesting an equivalence between a single daily dose and treatment conventional three daily doses.

OBJECTIVES The objective of this study is to verify the equivalence of using Clindamycin once a day versus 3 times daily in the rates of cure of septic abortion.

Hypotheses H0: Ps> Pn+2 The percentage of clinical cure with standard treatment (Ps) is greater than the rate of cure of alternative treatment + 2%.

Ha: Ps - 2% ≤ Pn The percentage of clinical cure with traditional treatment (Ps) minus 2% is less than or equal to the percentage of cure alternative treatment (Pn).

Variables

1. Standard treatment (Clindamycin 3x daily)
2. Alternative treatment (1x daily Clindamycin)
3. Clinical improvement (present or absent), defined as absence of fever (≤37.7 ° C), eating and walking without difficulty, as already described in the literature.

Materials and methods Design Randomized, prospective, double-blind study with two arms that follow the parameters of the CONSORT (17).

Geographic and temporal limitations The study will be conducted in patients attending the emergency unit at HCPA. A period of 24 months for data collection (about 4 patients per month), it will be necessary to reach sample size.

Inclusion criteria

All patients who come to emergency unit at HCPA with clinical diagnosis of septic abortion and will be treated with Clindamycin will be invited. The diagnosis of infected abortion is the same as used previously described by our group (9). Briefly, the presence of one of the criteria below in a < 20 weeks gestation, associated with a suspected ovular infection:

1. History of intrauterine manipulation with contaminated objects.
2. Vaginal discharge with foul odor.
3. Presence of pus flowing through the cervix.
4. Signs of peritoneal irritation.
5. leukocytosis (≥ 14,000 leukocytes / ml).
6. Warm Extremities, thready pulse and tachycardia (HR> 110 bpm)
7. Cyanosis and / or paleness
8. Tachypnea (MR> 30mrpm)
9. hypotension (Systolic Blood Pressure <90 mmHg)
10. Oliguria
11. Hyperthermia (≥ 37.8 ° C)

Exclusion criteria

Will be excluded all patients who:

1. Do not wish to participate in the project.
2. They used antibiotics prior to hospitalization (1 week period).
3. Being allergic to clindamycin or gentamicin.

Execution Patients eligible for the study will be invited to participate in the study at hospital admission for uterine curettage. After reading and signing the informed consent, patients will answer a standardized interview and after the interview, she will be randomized.

Randomization Subjects will be randomly allocated to treatment with clindamycin 3 times a day, or once a day; random sequence will be generated by a computer grouped into blocks of 4 treatments. The randomization sequence will be obtained from sequential sealed opaque envelope that will be in possession of the pharmacy emergency service HCPA. Researcher will not have access to the following treatment sequence. The Pharmacy Service will prepare the medication that will be part of routine emergency Gynecological Unit.

Patients and researchers will be blind to treatment allocation; saline infusion will be given in the place of clindamycin to keep patients blind to treatment arm.

Treatment

The regimen will consist of:

Standard treatment (Ps.): Clindamycin (900mg intravenously 8/8 hours diluted in 250 ml saline 0.9% solution (SF). The first vial of SF will contain 240 mg of gentamicin.

Alternative treatment (Pn): Clindamycin (2700mg) + gentamicin (240 mg) diluted in 250 ml of 0.9% saline. Two additional vials of SF 0.9% will be infused every 8 h as placebo.

The treatment will be continued up to 48 hours of good clinical condition, defined as absence of fever, decreased vaginal bleeding, minimal or no pain (AVS <4), eating, evacuating and walking normally.

Follow-up All women included in the study will be reviewed within 7 days after discharge as routine at the gynecologic emergency unit, to receive the results of the pathology.

Outcomes

The following outcomes will be assessed:

1. Clinical improvement until discharge in number of days of hospitalization, complications related to treatment.
2. Treatment failure will be considered as persistence of fever (≥37.8ºC) during hospital admission, worsening of abdominal pain, persistent vaginal bleeding, need for exchange clindamycin due to treatment failure, or the need to add other antibiotics, either intravenously or orally.
3. Hospital readmission within 7 days after discharge due to fever (Tax ≥37.8ºC), persistent pelvic pain, persistence or increase of uterine bleeding, or other hospital admission related to the septic abortion.
4. Presence of urinary tract infection or candidiasis will not be considered as treatment failure.

Sample Size The sample size was calculated as a trial of non-inferiority, using the formula proposed in the literature (18). According to data obtained in a retrospective study by our group (16) we expect that the estimated rate of clinical cure is 99% (95% CI - 95 to 99%) in the group with three daily doses and 100% (95% CI - 99 to 100%) in the experimental treatment. For a non-inferiority study, using a power of 90%, an alpha error of 5% and a lower limit for non-inferiority of 2%, 95 cases will be needed in each group.

Statistical analysis Data will be analyzed by intention to treat and per protocol. The definition of intention to treat is based on the criteria suggested in the literature. The statistical analysis will be performed using Student t-test to compare the difference of means; chi-square test will be used to compare proportions with confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Women with clinical diagnosis of septic abortion: Briefly, a suspicion of infected/septic abortion was confirmed by the presence of at least one of the following clinical signs: a history of intrauterine manipulation with contaminated objects; foul-smelling vaginal discharge; purulent discharge from the cervix; signs of peritoneal irritation; leukocytosis (leukocyte count > 14,000/mL); fever (temperature ≥ 37.8°C); or signs of a systemic inflammatory response, including tachycardia (heart rate > 110 bpm), tachypnoea (respiratory rate > 30 breaths/min), arterial hypotension (systolic blood pressure < 90 mmHg), oliguria, cyanosis, or pallor.

Exclusion Criteria:

* Refuse to participate in the study
* Use of antibiotics with 1 week prior randomization
* Known allergy to clindamycin or gentamycin

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 202 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized raw clinical data after completion of the study, through a URL
Supporting Information: SAP, Analytic Code
Time Frame: undefined
Access Criteria: public after completion, no access by now

REFERENCES:
- [Background] Singh S. Hospital admissions resulting from unsafe abortion: estimates from 13 developing countries. Lancet. 2006 Nov 25;368(9550):1887-92. doi: 10.1016/S0140-6736(06)69778-X. PMID 17126721
- [Background] Ahman E, Shah IH. New estimates and trends regarding unsafe abortion mortality. Int J Gynaecol Obstet. 2011 Nov;115(2):121-6. doi: 10.1016/j.ijgo.2011.05.027. Epub 2011 Aug 31. PMID 21885049
- [Background] Stubblefield PG, Grimes DA. Septic abortion. N Engl J Med. 1994 Aug 4;331(5):310-4. doi: 10.1056/NEJM199408043310507. PMID 8022443
- [Background] Del Priore G, Jackson-Stone M, Shim EK, Garfinkel J, Eichmann MA, Frederiksen MC. A comparison of once-daily and 8-hour gentamicin dosing in the treatment of postpartum endometritis. Obstet Gynecol. 1996 Jun;87(6):994-1000. doi: 10.1016/0029-7844(96)00054-3. PMID 8649712
- [Background] Hemsell DL, Martens MG, Faro S, Gall S, McGregor JA. A multicenter study comparing intravenous meropenem with clindamycin plus gentamicin for the treatment of acute gynecologic and obstetric pelvic infections in hospitalized women. Clin Infect Dis. 1997 Feb;24 Suppl 2:S222-30. doi: 10.1093/clinids/24.supplement_2.s222. PMID 9126697
- [Background] French LM, Smaill FM. Antibiotic regimens for endometritis after delivery. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD001067. doi: 10.1002/14651858.CD001067.pub2. PMID 15495005
- [Background] Savaris RF, de Moraes GS, Cristovam RA, Braun RD. Are antibiotics necessary after 48 hours of improvement in infected/septic abortions? A randomized controlled trial followed by a cohort study. Am J Obstet Gynecol. 2011 Apr;204(4):301.e1-5. doi: 10.1016/j.ajog.2010.11.017. Epub 2010 Dec 31. PMID 21195382
- [Background] Nicolau DP, Freeman CD, Belliveau PP, Nightingale CH, Ross JW, Quintiliani R. Experience with a once-daily aminoglycoside program administered to 2,184 adult patients. Antimicrob Agents Chemother. 1995 Mar;39(3):650-5. doi: 10.1128/AAC.39.3.650. PMID 7793867
- [Background] Rao SC, Srinivasjois R, Hagan R, Ahmed M. One dose per day compared to multiple doses per day of gentamicin for treatment of suspected or proven sepsis in neonates. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD005091. doi: 10.1002/14651858.CD005091.pub3. PMID 22071818
- [Background] Plaisance KI, Drusano GL, Forrest A, Townsend RJ, Standiford HC. Pharmacokinetic evaluation of two dosage regimens of clindamycin phosphate. Antimicrob Agents Chemother. 1989 May;33(5):618-20. doi: 10.1128/AAC.33.5.618. PMID 2751277
- [Background] Livingston JC, Llata E, Rinehart E, Leidwanger C, Mabie B, Haddad B, Sibai B. Gentamicin and clindamycin therapy in postpartum endometritis: the efficacy of daily dosing versus dosing every 8 hours. Am J Obstet Gynecol. 2003 Jan;188(1):149-52. doi: 10.1067/mob.2003.88. PMID 12548209
- [Background] Moberg PJ, Gottlieb C, Nord CE. Anaerobic bacteria in uterine infection following first trimester abortion. Eur J Clin Microbiol. 1982 Apr;1(2):82-6. doi: 10.1007/BF02014196. PMID 6890898
- [Background] Soper DE. Postpartum endometritis. Pathophysiology and prevention. J Reprod Med. 1988 Jan;33(1 Suppl):97-100. PMID 3278114
- [Background] Giugno CS, Silva AL, Fuhrich DG, Rabaioli PS, Goncalves KG, Sartor NC, Savaris RF. Daily dose of clindamycin versus standard divided doses in obstetrical and gynecological infections: a retrospective cohort study. Int J STD AIDS. 2013 Nov;24(11):893-8. doi: 10.1177/0956462413487516. Epub 2013 Jul 19. PMID 23970615
- [Background] Grimes DA. The "CONSORT" guidelines for randomized controlled trials in Obstetrics & Gynecology. Obstet Gynecol. 2002 Oct;100(4):631-2. doi: 10.1016/s0029-7844(02)02233-0. No abstract available. PMID 12383524
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between December 17, 2014, and December 31, 2023, at the gynecological emergency unit of Hospital de Clínicas de Porto Alegre, RS, Brazil.
Pre-assignment Details: Eligible patients will be invited to participate upon admission to the HCPA. After they read and sign the informed consent, patients will be randomized. Patients will be excluded from the study if they do not wish to participate, have used antimicrobials within one week of admission, or are allergic to clindamycin or gentamicin
Groups:
- clindamycin once a day: The intervention group received a single daily-dose regimen. At hour 0, participants were administered an infusion containing 240 mg of gentamicin and a total daily dose of 2700 mg of clindamycin. At hours 8 and 16, they received placebo infusions containing only the 0.9% saline solution.
- clindamycin thrice a day: The comparator group received the standard multiple-dose regimen. At hour 0, participants were administered an infusion containing 240 mg of gentamicin and 900 mg of clindamycin. At hours 8 and 16, they received subsequent infusions each containing 900 mg of clindamycin diluted in 250 ml bags of 0.9% saline solution
Period: Overall Study
Arm/Group | clindamycin once a day | clindamycin thrice a day
Started (Study was opened on December 4th, 2014) | 101 | 101
First enrolment (First enrolment for 3x/day was on Dec/17/2014. First enrolment for 1x/day was on Dec/24/2014.) | 1 | 1
Completed (Last participant 3x/day: Dec/12/2023 Last participant 1x/day: Dec/31/2023) | 101 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clindamycin Thrice a Day: Gentamycin 240mg i.v. once a day + plus clindamycin 900mg diluted in 250ml of sterile saline solution thrice a day.
- Total: Total of all reporting groups
Arm/Group | Clindamycin Once a Day | Clindamycin Thrice a Day | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] — age as a whole number
  years | 27.78 (7.72) | 29.11 (7.72) | 28.44 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants] — In total , we analyzed 202 participants for whom baseline characteristics were measured. In each arm, we had 101 participants and the entire study population was composed of women.
  Participants
    Female | 101 | 101 | 202
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 79 | 150
  Not Hispanic or Latino | 30 | 22 | 52
  Unknown or Not Reported | 0 | 0 | 0
Gestational age [Mean (Standard Deviation); unit: weeks] — gestational age measured in weeks and days
  weeks | 10.47 (4.09) | 10.74 (4.09) | 10.6 (4.15)

OUTCOME MEASURES:

1. Primary Outcome: Cure (Clinical Improvement Defined as Reduce of Pain, Bleeding and no Fever for 48h)
Description: Clinical improvement was defined by meeting all of the following criteria for a minimum of 48 consecutive hours: Reduction in pain, Reduction in vaginal bleeding, Absence of fever (afebrile)" Treatment failure was defined as the occurrence of any of the following events during hospital admission: Persistence of fever (temperature ≥37.8ºC), Worsening of abdominal pain, Persistent vaginal bleeding, Necessity to change the primary antibiotic (clindamycin), Addition of any other intravenous or oral antibiotics.
  For the purposes of analysis, patients who were lost to follow-up were classified as treatment failures.
Time Frame: cure at 72 hours
Population: no difference between values here and the numbers of participants, Intention To Treat
Measure: Number (95% Confidence Interval); unit: percentage of cure
Groups:
- clindamycin once a day: Clindamycin 2700mg+gentamicin 240mg+ 250ml sterile saline solution i.v. once a day until clinical improvement
- clindamycin thrice a day: Gentamycin 240mg i.v once a day, plus clindamycin 900mg i.v. 8/8 h diluted in 250ml of sterile saline solution
Arm/Group | clindamycin once a day | clindamycin thrice a day
Number analyzed (Participants) | 101 | 101
percentage of cure | 94.06 [87.64 to 97.25] | 86.14 [78.07 to 91.56]
Statistical Analysis 1: Comparison: clindamycin once a day vs clindamycin thrice a day; The null hypothesis (H₀) was that the treatment success rate of the once-daily clindamycin regimen is inferior to that of the thrice-daily regimen by a pre-specified non-inferiority margin (delta) of 2%. To achieve 90% power with a one-sided significance level (alpha) of 0.05 to reject the null hypothesis, a sample size of approximately 95 patients per group was required; Test type: Non-Inferiority — The non-inferiority margin was defined as a 2% difference. The sample size calculation aimed for 90% power at a 5% one-sided significance level, assuming clinical cure rates of 99% (standard arm) and 100% (experimental arm). This required 95 patients per arm, with a target enrollment of 100 per arm to account for potential dropouts; p = 0.06, Chi-squared; The 95% confidence interval for the difference in proportions between the two arms was calculated; Difference between 2 proportions = -0.02, 95% CI 1-sided [lower limit -0.02]

2. Secondary Outcome: Hospital Readmission Within 7 Days
Description: Number of patients who required hospital readmission for a repeat uterine curettage within 7 days of initial hospital discharge. Data was collected from patient's electronic medical records.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | clindamycin once a day | clindamycin thrice a day
Number analyzed (Participants) | 101 | 101
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: follow up within 7 days
Arm/Group | clindamycin once a day | clindamycin thrice a day
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/101
Other Adverse Events (participants affected / at risk) | 4/101 | 0/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | clindamycin once a day (N=101) | clindamycin thrice a day (N=101)
cutaneous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT02309346/Prot_SAP_000.pdf